CLINICAL TRIAL: NCT02109874
Title: A Phase I Randomized Placebo-Controlled, Double-Blind Study to Evaluate Safety and Immunogenicity of AERAS 404 When Administered as a Single Adjuvant Amount With Different Antigen Amounts in HIV-Negative BCG-Vaccinated Adults Without Evidence of Tuberculosis Infection
Brief Title: A Phase I Study to Evaluate Safety and Immunogenicity of AERAS 404 (C-011-404)
Acronym: C-011-404
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C-011-404
Record Dates: First submitted 2014-03-28; First posted 2014-04-10 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2014-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- AERAS-404 (mcg H4/nmol IC31) 5/500 (Experimental): H4 antigen (supplied in 4 different concentrations): 1.0 mL containing H4 antigen at 50, 150, 500, or 1500 mcg/mL in 10 mmol/L tris and 5% glycerol
  IC31 Adjuvant (supplied in 1 concentration): 0.8 mL containing IC31 adjuvant at 1250 nmol/mL, in 10 mmol/L tris and 169 mmol/L NaCl
  Interventions: Biological: AERAS-404 (mcg H4/nmol IC31)
- AERAS-404 (mcg H4/nmol IC31) 15/500 (Experimental): H4 antigen (supplied in 4 different concentrations): 1.0 mL containing H4 antigen at 50, 150, 500, or 1500 mcg/mL in 10 mmol/L tris and 5% glycerol
  IC31 Adjuvant (supplied in 1 concentration): 0.8 mL containing IC31 adjuvant at 1250 nmol/mL, in 10 mmol/L tris and 169 mmol/L NaCl
  Interventions: Biological: AERAS-404 (mcg H4/nmol IC31)
- AERAS-404 (mcg H4/nmol IC31) 50/500 (Experimental): H4 antigen (supplied in 4 different concentrations): 1.0 mL containing H4 antigen at 50, 150, 500, or 1500 mcg/mL in 10 mmol/L tris and 5% glycerol
  IC31 Adjuvant (supplied in 1 concentration): 0.8 mL containing IC31 adjuvant at 1250 nmol/mL, in 10 mmol/L tris and 169 mmol/L NaCl
  Interventions: Biological: AERAS-404 (mcg H4/nmol IC31)
- AERAS-404 (mcg H4/nmol IC31) 150/500 (Experimental): H4 antigen (supplied in 4 different concentrations): 1.0 mL containing H4 antigen at 50, 150, 500, or 1500 mcg/mL in 10 mmol/L tris and 5% glycerol
  IC31 Adjuvant (supplied in 1 concentration): 0.8 mL containing IC31 adjuvant at 1250 nmol/mL, in 10 mmol/L tris and 169 mmol/L NaCl
  Interventions: Biological: AERAS-404 (mcg H4/nmol IC31)
- Sterile buffer containing 10 mmol/L tris and 169 mmol/L NaCl (Placebo Comparator): Placebo: Sterile buffer containing 10 mmol/L tris and 169 mmol/L NaCl. This is the identical buffer solution in which IC31 is formulated.
  Interventions: Biological: Sterile buffer containing 10 mmol/L tris and 169 mmol/L NaCl

INTERVENTIONS:
Biological: AERAS-404 (mcg H4/nmol IC31) — Dose escalation
  Other Names: H4; AERAS-404
  Arms: AERAS-404 (mcg H4/nmol IC31) 15/500; AERAS-404 (mcg H4/nmol IC31) 150/500; AERAS-404 (mcg H4/nmol IC31) 5/500; AERAS-404 (mcg H4/nmol IC31) 50/500
Biological: Sterile buffer containing 10 mmol/L tris and 169 mmol/L NaCl
  Arms: Sterile buffer containing 10 mmol/L tris and 169 mmol/L NaCl

SUMMARY:
This Phase I study will be conducted as a randomized, placebo-controlled, double-blind, dose-escalation study in four groups of healthy adult male and female subjects who are BCG-vaccinated, HIV-negative, and have no evidence of tuberculosis infection. The study will be conducted at one or two sites located in South Africa. The purpose is to evaluate the safety and immunogenicity of two injections of AERAS 404 prepared with four escalating amounts of antigen in healthy adult male and female subjects who are BCG-vaccinated, HIV-negative, and have no evidence of tuberculosis infection.

DETAILED DESCRIPTION:
This Phase I study will be conducted as a randomized, placebo-controlled, double-blind, dose-escalation study in four groups of healthy adult male and female subjects who are BCG-vaccinated, HIV-negative, and have no evidence of tuberculosis infection. The study will be conducted at one or two sites located in South Africa.

Forty subjects will be sequentially enrolled into one of four study groups (i.e., Group 1, Group 2, Group 3, or Group 4) based on time of completion of screening, with 10 subjects enrolled into each group. Within each study group, subjects will be randomized to a treatment regimen of either AERAS-404 or placebo control administered by intramuscular injection on Study Day 0 and Study Day 56. All subjects will receive the same treatment on Study Day 0 as they receive on Study Day 56. The dose of antigen will increase between study groups. All subjects will be followed for safety and immunogenicity evaluations for 182 days. A total of eleven clinic visits are planned (excluding screening) for all subjects.

ELIGIBILITY:
Inclusion Criteria

Subjects must have met all of the following criteria:

1. Had completed written informed consent
2. Was male or female
3. Was age 18 through 50 years on Study Day 0
4. Had BCG vaccination at least 5 years ago, documented through medical history or presence of scar
5. Had general good health, confirmed by medical history and physical examination
6. Had a Body Mass Index (BMI) between 19 and 33 (weight in kg/[height in m]2)
7. Agreed to complete a follow-up period of 182 days as required by the protocol
8. Females: Agreed to avoid pregnancy from 28 days prior to Study Day 0 through the follow-up period of 182 days.
9. Agreed to avoid elective surgery for the duration of the study
10. Agreed to stay in contact with the investigative site for the duration of the study
11. Had completed simultaneous enrollment in Aeras Vaccine Development Registry protocol

Exclusion Criteria

Subjects must not have:

1. Acute illness on Study Day 0
2. Oral temperature equal to or greater than 37.5 degrees C on Study Day 0
3. Evidence of significant active infection
4. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted)
5. Received immunoglobulin or blood products within 42 days before Study Day 0
6. Received any investigational drug therapy or investigational vaccine within 182 days before Study Day 0
7. Received inactivated influenza vaccine or inactivated tick-borne encephalitis vaccine within 14 days before entry into the study, or any other standard vaccine within 42 days before Study Day 0 (the use of licensed drugs or vaccines medically indicated during the study interval was permitted)
8. Current chronic drug therapy including hormone replacement such as thyroxin, insulin, etc. Estrogen and progesterone replacement and contraceptives were acceptable.
9. History or laboratory evidence of any past, present or future possible immunodeficiency state which included (but was not limited to) any laboratory indication of HIV infection
10. History of allergic disease or reactions, including eczema, likely to be exacerbated by any component of the study vaccine
11. Previous medical history that may have compromised the safety of the subject in the study
12. Evidence of a new acute illness that may have compromised the safety of the subject in the study
13. Evidence of chronic hepatitis (e.g., hepatitis B core antibody or hepatitis C antibody)
14. Inability to discontinue daily medications except contraceptives during the study period
15. History of alcohol or drug abuse within the past 2 years
16. Tobacco or cannabis smoking 3 or more days per week
17. Positive urine test for illicit drugs (opiates, cocaine, amphetamines)
18. History or evidence of any systemic disease on physical examination or any acute or chronic illness that, in the opinion of the investigator, may have interfered with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy
19. History or evidence (including chest X-ray) of active tuberculosis
20. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
21. All females: Positive urine pregnancy test during screening; positive serum pregnancy test on the day of study vaccination; were nursing
22. Abnormal (per local laboratory parameters) chemistry, hematology or urinalysis obtained within 36 hours prior to randomization.
23. Laboratory evidence of Mtb infection, defined as a positive QuantiFERON-TB Gold (QFT-G) test.
24. History of a positive tuberculin skin test within the past ten years (defined according to local guidelines).
25. Received a tuberculin skin test within 3 months (90 days) prior to Study Day 0.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of two injections of AERAS 404 prepared with four escalating amounts of antigen in healthy adult subjects. Safety will be measured by number (percentage) and severity of SAEs. | Solicited and unsolicited AEs until study day 182
  The safety profile will be described by treatment regimen. Serious adverse events (SAE) will be collected on subjects throughout their participation in the study. Solicited and unsolicited adverse events will be captured for 28 days after each vaccination. The number (percentage) of subjects with any adverse events (including solicited, unsolicited and serious adverse events) will be summarized by MedRA system organ class (SOC) and preferred term (PT). Additional summaries will present the number (percentage) of subjects with any adverse events by severity and by relationship to study vaccine. The number (percentage) of subjects with post-vaccination clinical laboratory values or vital sign values recorded as newly abnormal following study vaccination and meeting toxicity criteria will be tabulated at each post-vaccination point and overall.

SECONDARY OUTCOMES:
Evaluate the immunogenicity of two injections of AERAS 404 prepared with four escalating amounts of antigen in healthy adult subjects. Immune response will be based on percentage of CD4+ and CD8+ cells. | 182 days
  The primary response will be measured by flow cytometry in the Intracellular cytokine staining (ICS) assay. Immune responses will be based on percentage of CD4+ and CD8+ T cells that produced one, two, or three cytokines (IFN-gamma, TNF, and/or IL-2) in response to stimulation with one of the 2 antigenic peptide pool (Ag85B and TB10.4) derived from and representing the entire amino acid sequences of teh mycobacterial antigens Ag85B and TB10.4.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkai Shi, MD, Study Director — Aeras
Locations (1):
- South African Tuberculosis Vaccine Institute; Brewelskloof Hospital, Worcester, South Africa

REFERENCES:
- [Background] Geldenhuys H, Mearns H, Miles DJ, Tameris M, Hokey D, Shi Z, Bennett S, Andersen P, Kromann I, Hoff ST, Hanekom WA, Mahomed H, Hatherill M, Scriba TJ; H4:IC31 Trial Study Group; van Rooyen M, Bruce McClain J, Ryall R, de Bruyn G; H4:IC31 Trial Study Groupa. The tuberculosis vaccine H4:IC31 is safe and induces a persistent polyfunctional CD4 T cell response in South African adults: A randomized controlled trial. Vaccine. 2015 Jul 9;33(30):3592-9. doi: 10.1016/j.vaccine.2015.05.036. Epub 2015 Jun 3. PMID 26048780